CLINICAL TRIAL: NCT03540238
Title: A Survey Investigating the Attitudes and Behaviors of Gastroenterology Specialists on Anesthesia Procedures in Endoscopy Units in Turkey
Brief Title: The Attitudes and Behaviors of Gastroenterology Specialists on Anesthesia Procedures in Endoscopy Units
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Ferda Yilmaz Inal, Assistant Professor, Istanbul Medeniyet University
Other Study IDs: 71306642-050.01.04
Record Dates: First submitted 2018-04-17; First posted 2018-05-30 (Actual); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Attitude, Staff; Behavior; Anesthesia
Keywords: sedation; endoscopy; anesthesia; gastroenterologist
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Most gastrointestinal endoscopic procedures are now performed with sedation and analgesia. Sedation and analgesia affects the quality of the procedure, patient co-operation and compliance as well as endoscopist's satisfaction. A wide variety of procedures have been reported worldwide for anesthesia during gastrointestinal endoscopy in adults.

The current survey was primarily designed to provide national data on the attidutes and behaviors of gastroentorologist on anesthesia procedures in endoscopy units in Turkey.

DETAILED DESCRIPTION:
Most gastrointestinal endoscopic procedures are now performed with sedation and analgesia. Sedation and analgesia affects the quality of the procedure, patient co-operation and compliance as well as endoscopist's satisfaction. Despite the use of numerous sedation and analgesic techniques for GI endoscopy procedures, the best method is still controversial. A wide variety of procedures have been reported worldwide for anesthesia during gastrointestinal endoscopy in adults.The current survey was primarily designed to provide national data on current sedation and monitoring practices that was carried out during gastrointestinal endoscopy. Secondary objectives were to provide data on the endoscopic application of the turkish gastroenterologist.

The questionnaire consisting of 20 questions about the anesthesia methods applied in the procedures in the endoscopy unit will be sent to 1000 gastroenterologists registered in the Turkish Gastroenterology Association by e-mail. The questionnaire is covered the demographic data, types of endoscopic procedures and anesthesia methods applied, anesthetic agents, monitoring methods, anesthesia team, preanesthetic evaluation and consent forms, recovery unit and complications and interventions during anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Being a Gastroenterology specialist

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Active working gastrology specialist
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2018-05-16 (Actual); Primary Completion 2018-06-15 (Estimated); Study Completion 2018-06-15 (Estimated)

PRIMARY OUTCOMES:
gastroenterology specialists' anesthesia choices | 1 day
  questions to know their current anesthesia and monitoring practices during endoscopic procedures

CONTACTS AND LOCATIONS:
Locations (1):
- Ferda Yılmaz Inal, Istanbul, Turkey (Türkiye)